CLINICAL TRIAL: NCT00504400
Title: Ranibizumab in Idiopathic Macular Telangiectasia, Type 2. A Prospective Interventional Non-randomized Study Comparing the Efficacy and Safety of Intravitreal Ranibizumab in Type 2 Idiopathic Macular Telangiectasia.
Brief Title: Ranibizumab to Treat Type 2 Idiopathic Macular Telangiectasia (RAMA-Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Novartis (Industry)
Responsible Party: University of Bonn, University of Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002ADE04; EudraCT number 2006-006233-40
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Idiopathic Macular Telangiectasia
Keywords: macular telangiectasia; parafoveal telangiectasis; nonproliferative; therapy; intravitreal injection; ranibizumab; lucentis
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Intravitreal injection ranibizumab

INTERVENTIONS:
Drug: Intravitreal injection ranibizumab — Monthly intravitreal injection of of 0.5mg ranibizumab in one eye over one year
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to investigate if a new drug called ranibizumab is effective to treat a rare bilateral disease of the macula: type 2 idiopathic macular telangiectasia (type 2 IMT). 10 patients will receive monthly injections of the drug into one eye over a period of one year.

DETAILED DESCRIPTION:
Type 2 idiopathic macular telangiectasia (type 2 IMT) is a retinal disease of unknown etiology that commonly presents with a slow decrease in visual acuity, reading difficulties and metamorphopsia in the fifth to seventh decade. Diagnosis is based on fluorescein angiography which typically reveals parafoveal leakage in the late phase and may show telangiectatic capillaries in the early phase. In a subset of patients, a proliferative stage with secondary neovascularizations may develop late in the disease course. In the past, there has been no effective treatment for the disease stages without neovascularization.

Recent studies in a limited number of patients with nonproliferative disease have shown promising results after intravitreal injection of bevacizumab, an antagonist targeting vascular endothelial growth factor (VEGF). Bevacizumab resulted in a decrease of parafoveal leakage in fluorescein angiography and a decrease in retinal thickness. An increase in visual acuity was reported in a subset of patients.

The RAMA-Trial is initiated in order to investigate the effect of a ranibizumab. The safety and tolerability of this VEGF-antagonist has been extensively studied in large cohorts of patients suffering from age-related macular degeneration.

Patients with type 2 IMT will receive monthly injections over a period of one year. The above mentioned outcome measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 idiopathic macular telangiectasia
* minimum of 18 years
* patient must be able to follow protocol
* written informed consent
* best corrected visual acuity between 20/200 - 20/32 in the treated eye

Exclusion Criteria:

* patients who do not fulfill the inclusion criteria
* patients with other retinal vascular disease such as diabetic retinopathy or venous occlusive diseases
* ocular surgery 3 months before study enrollment
* history of uncontrolled glaucoma
* active intraocular inflammation or inflammation of the ocular adnexa
* subfoveal fibrosis in the study eye
* inability to follow study protocol
* major surgery one month before study enrollment
* history of severe cardiovascular disease or history of stroke 6 months before study enrollment
* allergies against substances or components of the study medication
* low anticipated compliance
* patients who participate(d) in clinical trials simultaneously or within the last 60 days
* pregnancy, lactation, women that may become pregnant and don't use safe contraception
* chronic alcohol- or drug abuse within the last year
* lacking legal competence or language ability
* neurologic diseases such as multiple sclerosis
* need of concomitant medication that is not allowed in combination with ranibizumab
* previous intravitreal therapy with anti-angiogenic substances in the study eye within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | one year

SECONDARY OUTCOMES:
Reading ability | one year
Scotomas measured by means of microperimetry | one year
Changes in retinal thickness assessed by optical coherence tomography (OCT) imaging | one year
Changes in parafoveal leakage assessed by fluorescein angiography | one year
Quality of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Frank Holz, MD, Principal Investigator — University of Bonn, Department of Ophthalmology; Hendrik PN Scholl, MD, MA, Principal Investigator — University of Bonn
Locations (1):
- Department of Ophthalmology, University of Bonn, Bonn, Germany

REFERENCES:
- [Derived] Charbel Issa P, Finger RP, Kruse K, Baumuller S, Scholl HP, Holz FG. Monthly ranibizumab for nonproliferative macular telangiectasia type 2: a 12-month prospective study. Am J Ophthalmol. 2011 May;151(5):876-886.e1. doi: 10.1016/j.ajo.2010.11.019. Epub 2011 Feb 19. PMID 21334595
- [Derived] Charbel Issa P, Troeger E, Finger R, Holz FG, Wilke R, Scholl HP. Structure-function correlation of the human central retina. PLoS One. 2010 Sep 22;5(9):e12864. doi: 10.1371/journal.pone.0012864. PMID 20877651
- See also: Related Info — http://www.augenklinik.uni-bonn.de